CLINICAL TRIAL: NCT03300271
Title: Effects of a Supportive Mobile Health for Life Style Modification on Blood Pressure and Insulin Resistance Improvement in People With Metabolic Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2017-0666
Record Dates: First submitted 2017-09-24; First posted 2017-10-03 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the experimental conditions (mobile application), or the usual condition (education).
Who Masked: Investigator, Outcomes Assessor
Masking Description: A designated researcher will be responsible for the random allocation and mask the results, so the investigators and the outcomes assessor do know the which group the participants are been allocated in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No intervention (Education) (Other): Participants in this group is provided education. Education includes information of metabolic syndrome, methods to manage lifestyle (diet, physical activity).
  Interventions: Other: Education
- Mobile Application (Self monitoring) (Experimental): Participants in this group will be introduced to use a mobile application to self record and monitor their life style behaviors. They will be also be provided education same as the control group.
  Interventions: Other: Mobile application for self monitoring
- Mobile Application (Personal coaching) (Experimental): Participants in this group will be introduced to use a mobile application. Personal coaches such as dietitian, sports manager encourage to improve their life style behaviors. They will be also be provided education same as the control group.
  Interventions: Other: Mobile application for personal coaching

INTERVENTIONS:
Other: Mobile application for self monitoring — Participants in this group will be introduced to use a mobile application to self record and monitor their life style behaviors. They will be also be provided education same as the control group.
  Arms: Mobile Application (Self monitoring)
Other: Education — Participants in this group is provided education. Education includes information of metabolic syndrome, methods to manage lifestyle (diet, physical activity).
  Arms: No intervention (Education)
Other: Mobile application for personal coaching — Participants in this group will be introduced to use a mobile application. Personal coaches such as dietitian, sports manager encourage to improve their life style behaviors. They will be also be provided education same as the control group.
  Arms: Mobile Application (Personal coaching)

SUMMARY:
The purpose of this randomized study is to assess the efficacy of a mobile application for the improvement of blood pressure and insulin resistance in people with metabolic abnormalities.

DETAILED DESCRIPTION:
The purpose of this randomized study is to assess the efficacy of a mobile application for the improvement of blood pressure and insulin resistance in people with metabolic syndrome.

This study is a 24 week follow up randomized prevention trial. Participants visit for a screening test, then eligible participants are randomly assigned for one of the following arms; 1 intervention group using a mobile application to monitor their life style behaviors, 1 intervention group using a mobile application for personal coaching on purpose of improving their life style behavior, and 1 control group providing education about managing life style behaviors.

ELIGIBILITY:
Inclusion Criteria:

* "Etiologic study on cardiovascular and metabolic diseases: prospective cohort study (Severance Hospital IRB No. 4-2013-0661)" participants
* Smartphone user
* Metabolic abnormality. Having 2 or more components of metabolic syndrome described below:

  1. Central obesity : waist circumference ≥ 90cm in male, ≥ 80cm in female
  2. Systolic/diastolic blood pressure ≥ 130/85 mmHg
  3. Serum triglyceride ≥ 150 mg/dL
  4. Serum high density lipoprotein cholesterol < 40 mg/dL in male, 50 mg/dL in female
  5. Fasting glucose ≥ 100mg/dL

Exclusion Criteria:

* Presently or planning for pregnant/breastfeeding during the study. Or confirmed pregnancy by a urine test.
* Currently taking medication (including insulin injection) for hypertension, dyslipidemia, or diabetes.
* Presently using a mobile application for lifestyle modification

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Change in systolic/diastolic blood pressures | 24 weeks
  Change of systolic/diastolic blood pressures and insulin resistance are the differences between the last visit and baseline (screening visit).

SECONDARY OUTCOMES:
Change in the eligibility criteria for metabolic syndrome | 24 weeks
  Change of metabolic profiles are the differences between the last visit and baseline (screening visit).

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho SMJ, Lee JH, Shim JS, Yeom H, Lee SJ, Jeon YW, Kim HC. Effect of Smartphone-Based Lifestyle Coaching App on Community-Dwelling Population With Moderate Metabolic Abnormalities: Randomized Controlled Trial. J Med Internet Res. 2020 Oct 9;22(10):e17435. doi: 10.2196/17435. PMID 33034564